CLINICAL TRIAL: NCT02360176
Title: Evaluation of Minimally Invasive Bariatric Surgery Using a Single Laparoscopic Trocar (Single Incision of 2.5 to 3 cm) Versus 4 to 7 Trocars in Sleeve Gastrectomy
Brief Title: Benefit of Single Port-surgery in Sleeve Gastrectomy
Acronym: MINIOB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130940
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Surgical Treatment of Obesity
Keywords: single port surgery; bariatric surgery; sleeve gastrectomy; randomise prospective study; complication rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleeve gastrectomy single port (Experimental): Sleeve gastrectomy single port
  Interventions: Procedure: Sleeve gastrectomy single port
- Sleeve gastrectomy multi trocar (Active Comparator): Sleeve gastrectomy multi trocar
  Interventions: Procedure: Sleeve gastrectomy multi trocar

INTERVENTIONS:
Procedure: Sleeve gastrectomy single port — Bariatric surgery: one incision of 2.5 to 3 cm
  Arms: Sleeve gastrectomy single port
Procedure: Sleeve gastrectomy multi trocar — Bariatric surgery: 4 to 7 incisions of 1 to 2 cm
  Arms: Sleeve gastrectomy multi trocar

SUMMARY:
Demonstrate non-inferiority of the single port for sleeve gastrectomy compared to the reference method in terms of complications using a score of morbidity and mortality at 6 and 24 months: Rate of fistula, intra and extra abdominal abcess, hemorrhage, gastric stenosis, splenic lesions, hernia, residual gastric pouch and mortality

DETAILED DESCRIPTION:
The single port surgery is the natural evolution of laparoscopy. To date only few studies have evaluated the feasibility of this technique in sleeve gastrectomy. The investigators want to demonstrate the non-inferiority in terms of morbidity-mortality of use single trocar in sleeve gastrectomy compared the multiport technique. Moreover it should highlight the non-inferiority in terms of anatomical quality, reduction of excess weight lost, reduction of comorbidities, decrease post operative pain, improved quality of life and evaluate medico-economic impact of these technique to validating this new surgical approach for bariatric surgery. The study will be multicentric with 6 university center (Montpellier, Amiens, Lille, Creteil, Poissy and Montsouris Institut). 388 patients will be included in the tow group of the prospective randomise study.

ELIGIBILITY:
Inclusion Criteria:

* BMI> 35 kg/m2 with comorbidity (s) or> 40 kg/m2
* Patients aged 18 to 65 years
* Discussion and decision sleeve gastrectomy multidisciplinary meeting
* Free, informed and written consent
* Affiliation to a social security or other assurance

Exclusion Criteria - Anesthetics

Exclusion Criteria:

* Uncontrolled severe infection
* Liver disease other than obesity pathology
* Pregnancy (positive hCG)
* Large hiatal hernia
* Esophagitis uncontrolled
* History of gastric bypass and gastric surgery other than gastric banding
* Saving Justice guardianship
* Participation in another ongoing study
* Cognitive or severe mental illness
* Severe and non-stabilized eating disorders
* Addiction to alcohol and psychoactive substances"

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Complication rate | up to 24 months
  The principal criteria of analysis will be a score of morbidity and mortality at 24 months including: rate of fistula and intra-abdominal abscesses, the bleeding rate, the rate of gastric stenosis, rate splenic lesions, residual pouch or parietal damage (abscesses, incisional hernia, hematoma, delayed wound healing), and death

SECONDARY OUTCOMES:
Complication rate | up 3, 6, 9, and 12 months
Reduction of excess weight by measuring BMI in kg / m2 pre-and postoperatively | up 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pourcher, MD PhD, Principal Investigator — Montsouris Institut
Locations (1):
- Montsouris Insitut, Paris, France

IPD SHARING:
Plan to Share IPD: No